CLINICAL TRIAL: NCT06709014
Title: A 6-month & 18-month Prospective, Randomized, Placebo-controlled, Double-blind Dual Clinical Trial Investigating Efficacy and Safety of Buntanetap in Treating Participants of Early Alzheimer's Disease
Brief Title: A Double-blind Dual Study Assessing Safety and Efficacy of Buntanetap in Participants With Early AD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Collaborators: Prevail Infoworks (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANVS-25001
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-04

CONDITIONS: Early Alzheimers Disease
Keywords: Early Alzheimers disease; Early AD; AD; mild cognitive impairment; MCI; buntanetap; posiphen
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — phenserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study partner will also be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- buntanetap (Experimental)
  Interventions: Drug: buntanetap/posiphen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: buntanetap/posiphen — 30mg capsule by mouth once daily for 18 months
  Arms: buntanetap
Drug: Placebo — Placebo capsule by mouth once daily for 18 months
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if buntanetap/Posiphen works to treat early Alzheimer's disease in adults aged 55-85. It will also learn about the safety of buntanetap/Posiphen. The main questions it aims to answer are:

* Does buntanetap/Posiphen improve cognition as measured by ADAS-Cog13?
* Does buntanetap/Posiphen improve function as measured by ADCS-iADL?
* What medical issues do participants have, if any, when taking buntanetap/Posiphen?

Researchers will compare buntanetap/Posiphen to a placebo (a look-alike substance that contains no drug) to see if buntanetap/Posiphen works to treat early Alzheimer's disease.

Participants will:

* Take buntanetap/Posiphen or a placebo every day for 18 months
* Visit the clinic periodically for checkups, tests, and questionnaires (screening visits, enrollment, month 1, month 3, month 6, month 9, month 12, month 15, month 18), including a volumetric MRI at month 6 and month 18
* Complete pre- and post-clinic visit phone calls

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AD according to the 2024 National Institute on Aging and Alzheimer's Association criteria.
2. Male or female, aged 55 - 85 years.
3. MMSE 20-28 at screening and baseline.
4. CDR global score=0.5 or 1, with memory box score at least 0.5 at screening and baseline.
5. Positive for amyloid beta as defined by plasma p-tau217 level at screening.
6. Neuroimaging (MRI) consistent with the clinical diagnosis of AD and without findings of significant exclusionary abnormalities (see exclusion criteria # 4). A historical MRI, up to 1 year prior to screening, may be used as long as there have been no interval clinical neurologic events that may suggest a change in the MRI scan.
7. Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week) and will accompany the participant on study visits at designated times.
8. Female participants of childbearing potential* must have a negative urine pregnancy test at screening, must be non-lactating and must agree to use a highly effective method of contraception (i.e., a method resulting in a failure rate of less than 1% per year when used consistently and correctly) during the trial and for one month after the last dose of trial treatment, such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation,
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation,
   * Intrauterine device (IUD),
   * Intrauterine hormone-releasing system (IUS),
   * Bilateral tubal occlusion,
   * Vasectomized partner (a vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the participant. If not, an additional highly effective method of contraception should be used),
   * Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant).

     * Non-childbearing potential includes surgically sterilized or postmenopausal with no menstrual bleeding for at least one year prior to study start.
9. Male participants must be sterile or sexually inactive or agree not to father a child during the study and one month after the last dose of study medication and must agree to use a barrier method for contraception. Female partners of male participants must adopt a highly effective method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation,
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation,
   * IUD,
   * IUS,
   * Bilateral tubal occlusion.
10. General cognition and functional performance sufficiently preserved that the subject can provide written informed consent. At re-consent, a legally authorized representative may co-sign if participants do not meet the general cognition and functional performance needed in the opinion of the investigator.
11. No evidence of current suicidal ideation or previous suicide attempt in the past month as evaluated in the Columbia Suicide Severity Rating Scale.
12. Stability of permitted medications for at least 4 weeks prior to screening. Refer to Concomitant Medications section for details on prohibited and permitted medications.

    * Cholinesterase inhibitors and/or memantine medication,
    * Anticonvulsant medications used for epilepsy or mood stabilization, or neuropathic pain indications, and have not had a breakthrough seizure in 3 years prior to screening
    * Mood-stabilizing psychotropic agents including, but not limited to, lithium.
13. Adequate visual and hearing ability (physical ability to perform all the study assessments).
14. Participants previously exposed to buntanetap can still be included in the study after a 28-day wash out period.

Exclusion Criteria:

1. Has a history of psychiatric disorder such as schizophrenia, bipolar disorder, or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM), unless they are stable on treatment or no longer need treatment. Mild depression or history of depression that is stable on treatment with selective serotonin reuptake inhibitors (SSRI), serotonin and norepinephrine reuptake inhibitors (SNRI) or other anti-depression medication (e.g. Wellbutrin) at a stable dose is acceptable. Refer to Concomitant Medications section above for details on prohibited and permitted medications.
2. Has non-AD dementia, such as vascular dementia, Lewy body dementia, frontotemporal disease, PD dementia, B12 and thyroid deficiency caused dementia.
3. History of a seizure disorder, if stable on medication is acceptable. Refer to Concomitant Medications section above for details on prohibited and permitted medications.
4. Screening MRI (or historical MRI, if applicable) of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage (>5) or infarct > 1 cm3, > 3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g., abscess or brain tumor such as meningioma unless they are documented and stable).
5. Has a history or current evidence of long QT syndrome, Fridericia's formula corrected QT (QTcF) interval ≥ 450 ms for men and ≥ 460 ms for women ((in the absence of a bundle branch block), or torsades de pointes.
6. Has bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG at screening and deemed medically significant by the PI.
7. Has uncontrolled Type-1 or Type-2 diabetes. A participant with hemoglobin subunit alpha 1c (HbA1c) levels up to 7.5% can be enrolled if the PI believes the participant's diabetes is under control.
8. Has clinically significant renal (Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) <50 mL/min/BSA (body surface area) or hepatic impairment (alkaline phosphatase (ALP) > 2.0 ULN and/or total bilirubin > 2.0 ULN).
9. Has any clinically significant abnormal laboratory values. Participants with liver function tests (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) greater than twice the upper limit of normal will be excluded.
10. Is at imminent risk of self-harm, based on clinical interview and responses on the C- SSRS, or of harm to others in the opinion of the PI. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or method (e.g., positive response to items 4 or 5 in assessment of suicidal ideation on the C-SSRS) in the past 2 months, or suicidal behavior in the past 6 months.
11. Has cancer or has had a malignant tumor within the past year, except participants who underwent potentially curative therapy with no evidence of recurrence (participants with stable untreated cancer are not excluded).
12. Alcohol / Substance use disorder, moderate to severe, in the last 5 years according to the most current version DSM.
13. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 4 weeks prior to the start of screening, or five half-lives of the investigational drug, whichever is greater. The end of a previous investigational trial is the date the last dose of an investigational agent was taken.
14. Participants with learning disability or developmental delay.
15. Participants whom the PI deems to be otherwise ineligible.
16. Participants with a known allergy to the investigational drug or any of its components.

    Inactive ingredients of the investigational medicinal product:
    * Silicified Microcrystalline Cellulose
    * Dibasic Calcium Phosphate Dihydrate
    * Mannitol
    * Stearic Acid
    * Hypromellosee (capsule shells structure)
    * Titanium dioxide (opacifier of the capsule shells)
17. Participant is currently pregnant, breast-feeding, and/or lactating.
18. Participant is currently taking strong and moderate CYP3A4 inhibitors and/or inducers. Refer to Concomitant Medications section below for details on prohibited and permitted medications.
19. Participants with uncontrolled hypertension (systolic >160mm Hg and/or diastolic >95mm Hg) or hypotension (systolic <90mm Hg and/or diastolic <60 mm Hg) and deemed medically significant by the PI.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale 13 (ADAS-Cog13) | From screening to 6-month readout, to end of treatment at 18 months.
  ADAS-Cog13 includes the original ADAS-Cog11 items that assess cognitive function across the memory, language, praxis, and orientation domains and adds a number cancellation task and a delayed free recall task. Total scores range from 0-85, with higher scores indicating greater cognitive impairment.
Alzheimer's Disease Cooperative Study-Instrumental Activities of Daily Living Scale (ADCS-iADL) | From screening to 6-month readout, to end of treatment at 18 months.
  The Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale (ADCS-ADL) is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's study partner to assess function to the degree to which the participant can perform a variety of tasks. The questionnaire asks 6 questions of basic ADLs and 17 instrumental ADLs. The iADL are more complex tasks, including activities such as shopping, maintaining appointments, or managing one's belongings or finances. The ADCS-iADL subset is assessed with items 6a and 7-23; scores range from 0 to 59, with lower scores indicating greater impairment in function.

CONTACTS AND LOCATIONS:
Locations (83):
- United States (83):
  - MD First Research, Chandler, Arizona
  - Xenoscience, Phoenix, Arizona
  - Clinical Endpoints, Scottsdale, Arizona
  - Advanced Research Center, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - Eximia Clinical Research, Encino, California
  - Sun Valley Research, Imperial, California
  - Mary S. Easton Center for Alzheimer's Research and Care, UCLA, Los Angeles, California
  - UC Davis Alzheimer's Disease Research Center, Sacramento, California
  - The Neuron Clinic, San Marcos, California
  - Mountain Neurological Center, Basalt, Colorado
  - CenExel Rocky Mountain, Englewood, Colorado
  - Research Center for Clinical Trials, Norwalk, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - SFM Clinical Research, Boca Raton, Florida
  - K2 Medical Research, Clermont, Florida
  - K2 Medical Research Daytona, Daytona Beach, Florida
  - Neuropsychiatric Research Center, Fort Myers, Florida
  - Velocity Clinical, Hallandale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - K2 Medical Research, Lady Lake, Florida
  - Headlands Research JEM, Lake Worth, Florida
  - Accel Research Sites Lakeland (Alcanza), Lakeland, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud Clinical Research, Melbourne, Florida
  - Flourish Research/Merritt Island Medical Research, Merritt Island, Florida
  - Miami Jewish Health, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Conquest Research, Orlando, Florida
  - Axiom Brain Health, LLC, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - Accel Neurosciences, Decatur, Georgia
  - CARE (Center for Advanced Research & Education), Gainesville, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Re:Cognition Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Charter Research Chicago, Chicago, Illinois
  - Great Lakes Clinical Trials/Flourish Research, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - JWM Research, Indianaopolis, Indiana
  - Ascension via Christi Research, Wichita, Kansas
  - Tandem Intermediate, Metairie, Louisiana
  - Headlands Research Pharmasite, Pikesville, Maryland
  - Neurology Center of New England, PC, Foxborough, Massachusetts
  - Headlands Research Easter Massachusetts, Plymouth, Massachusetts
  - Mayflower Clinical, Russells Mills, Massachusetts
  - Elixia MA, Springfield, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Precise Research Center, Flowood, Mississippi
  - Clinical Research Professionals - Headlands Research, Chesterfield, Missouri
  - Oasis Clinical Trials LLC, Las Vegas, Nevada
  - Cenexel Advanced Medical Research of New Jersey (AMRI), Toms River, New Jersey
  - Advanced Clinical Institute, West Long Branch, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - SPRI, Brooklyn, New York
  - Neurological Associates of Long Island, Lake Success, New York
  - Parker Jewish Institute for Health Care and Rehab, New Hyde Park, New York
  - New York Neurology Associates, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Ichor Research, Syracuse, New York
  - Duke University, Durham, North Carolina
  - AMC Research/Flourish Research, Matthews, North Carolina
  - Eximia Clinical Research, Raleigh, North Carolina
  - American Clinical Research Center, Beavercreek, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Insight Clinical Trials, Independence, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Summit Headlands, Portland, Oregon
  - Abington Neurologic Associates, Abington, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - K2 Keystone, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Palmetto Primary Care & Specialty Physicians, Summerville, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - K2 Medical Research Nashville, Nashville, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - NeuroMind Clinical Trials, Houston, Texas
  - Central Texas Neurology Associates, Round Rock, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Memory Clinic, Inc., Bennington, Vermont
  - Sana Research, Arlington, Virginia
  - Re:Cognition Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Annovis Bio website — https://www.annovisbio.com/